CLINICAL TRIAL: NCT01641549
Title: Surgery Compared to Fibrinolytic Therapy for Symptomatic Patients With Left-sided Prosthetic Heart Valve Thrombosis
Brief Title: Surgery Versus Fibrinolytic Therapy for Left-sided Prosthetic Heart Valve Thrombosis
Acronym: SAFE-PVT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Ganesan Karthikeyan, Additional Professor of Cardiology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 1.01
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Left-sided Prosthetic Heart Valve Thrombosis
Keywords: Prosthetic valve thrombosis; Fibrinolytic therapy; Emergency surgery
MeSH Terms: interventions — Thrombolytic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emergency surgery (Experimental): Emergency surgery (valve replacement or thrombectomy)
  Interventions: Procedure: Emergency surgery
- Fibrinolytic therapy (Active Comparator): Streptokinase (SK) at a dose of 0.25MU over 30 minutes followed by a 0.1MU/ hour infusion, or other fibrinolytic agent
  Interventions: Drug: Fibrinolytic therapy

INTERVENTIONS:
Procedure: Emergency surgery — Emergency surgery (valve replacement or thrombectomy)
  Other Names: Redo valve replacement
  Arms: Emergency surgery
Drug: Fibrinolytic therapy — Streptokinase (SK) at a dose of 0.25MU over 30 minutes followed by a 0.1MU/ hour infusion, or other fibrinolytic agent at standard doses
  Other Names: Thrombolytic therapy
  Arms: Fibrinolytic therapy

SUMMARY:
Malfunction of mechanical heart valves due to clot formation is a potentially devastating complication. It often results in heart failure, death or stroke. This condition occurs frequently in patients with mechanical valves in developing countries because they are unable to monitor and adjust the dose of blood thinning medications. The best treatment modality for the treatment of patients with this condition is not known. There is no reliable data from clinical trials to guide treatment and there are no firm guidelines. Treatment with clot-busting drugs is most commonly used because these drugs (e.g., streptokinase) are readily available, cheap, and easy to use. However, this treatment is associated with high rates of treatment-related side-effects (death, life-threatening bleeding and stroke). Moreover, some recent studies suggest that clot-busting drugs may not be as efficacious in restoring valve function, as previously believed. Emergency surgery is less often used because it is more expensive and the required facilities and manpower are not available at all times at all places. But there is evidence to suggest that surgery results in better success rates with a lower risk of bleeding and stroke. Well-designed prospective randomised trials (the "gold-standard" for reliable evidence) comparing the efficacy, safety and cost-effectiveness of the two modalities, are needed to help doctors in developing countries make informed decisions when treating patients with clotted mechanical heart valves. The investigators propose to perform a randomised controlled trial comparing emergency surgery with treatment with clot-busting agents in patients with clotted mechanical valves. The study will be conducted over 4 years at a single, university hospital in a developing country. This study will determine how often patients who are treated with surgery will be discharged from hospital, with completely restored valve function, without having suffered a stroke or life-threatening bleeding, when compared to those who received clot-busting drugs. The investigators will also find out which of the treatments is safe and cost-effective.

DETAILED DESCRIPTION:
Left-sided prosthetic valve thrombosis (PVT) is a potentially devastating complication which can affect patients with mechanical heart valves. It occurs frequently in developing countries because of poor anticoagulation quality. The best modality for treating this condition is not known. Most of the available data is from retrospective studies and case series, and current guidelines are based largely on expert opinion. Therefore recommendations for treatment vary widely. Fibrinolytic therapy (FT) is the most commonly used treatment because fibrinolytic agents such as streptokinase are readily available, cheap, and easy to use. However, FT is associated with high rates of treatment-related adverse effects (death, major bleeding and stroke). Moreover, recent studies suggest that FT may not be as efficacious in restoring valve function, as previously believed. Emergency surgery is less often used because it is more expensive and the required facilities and manpower are not available at all times at all places. A systematic review and meta-analysis of the available literature that the investigators performed, suggests that surgery may result in better success rates with a lower risk of major bleeding, stroke and non-CNS systemic embolism. Evidence from well designed randomised controlled trials is needed to determine the optimal treatment of left-sided PVT. The investigators propose to do a single-centre, open-label, randomised controlled trial comparing emergency surgery with FT for the treatment of symptomatic patients with left-sided PVT. The primary outcome is the occurrence of a complete clinical response, defined as discharge from hospital with completely restored valve function, in the absence of stroke, major bleeding or non-CNS systemic embolism. The investigators will compare the safety of the two interventions and quality of life at discharge and at 1 year. The investigators will also assess the cost-effectiveness of surgery compared to FT from a societal perspective in the context of the Indian healthcare system

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age with recent-onset (≤2 weeks), objectively diagnosed, symptomatic (NYHA class II-IV) left-sided prosthetic valve dysfunction

Exclusion Criteria:

* Absolute contraindications to FT (any history of intracranial hemorrhage, active bleeding from any site, ischemic stroke in the preceding 3 months, left atrial thrombus on TTE)
* Pregnant patients
* Asymptomatic patients (incidentally detected valve thrombosis)
* Inability to obtain (or refusal to provide) informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response | In-hospital, average of 10 days
  The primary outcome is the occurrence of a complete clinical response, defined as discharge from hospital with completely restored valve function, in the absence of stroke, major bleeding or non-CNS systemic embolism.

SECONDARY OUTCOMES:
Death, stroke, major bleeding, or non-CNS systemic embolism | In-hospital, average of 10 days
  A composite of in-hospital death, stroke, major bleeding or non-CNS systemic embolism.
Death, recurrent PVT, stroke or non-CNS systemic embolism or persistent abnormal valve function | 1 year
  A composite of death, recurrent PVT, stroke or non-CNS systemic embolism, and persistent abnormal valve function (or re-do surgery for persistent valve dysfunction)

CONTACTS AND LOCATIONS:
Overall Officials: Ganesan Karthikeyan, MD, DM, MSc, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Departments of cardiology and Cardiovascular Surgery, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided